CLINICAL TRIAL: NCT00801866
Title: Prevention of Post-photocoagulation Macular Edema by Intravitreal Bevacizumab.
Brief Title: Avastin for Post-photocoagulation Macular Edema
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: undefined
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: APEC-035
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Macular Edema
Keywords: Panretinal Photocoagulation; Macular Edema; Intravitreal Bevacizumab
MeSH Terms: conditions — Macular Edema | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Panretinal Photocoagulation + Bevacizumab
  Interventions: Drug: Bevacizumab
- Group 2 (Experimental): Panretinal Photocoagulation
  Interventions: Procedure: Panretinal Photocoagulation

INTERVENTIONS:
Drug: Bevacizumab — Intravitreal administration
  Arms: Group 1
Procedure: Panretinal Photocoagulation — Panretinal Photocoagulation
  Arms: Group 2

SUMMARY:
to evaluate the efficacy of a single intravitreal bevacizumab (IVB) injection, 0.1mL (2.5mg), against panretinal photocoagulation (PRP)-induced macular thickening and visual disturbance in patients with severe nonproliferative diabetic retinopathy (NPDR) and proliferative diabetic retinopathy (PDR) and good vision

ELIGIBILITY:
Inclusion Criteria:

* Patients with Proliferative retinopathy or severe non-proliferative retinopathy
* BCVA of 20/63 or better (56 ETDRS letters
* No history of Macular Edema
* Central Retinal Thickness of 250mics or more

Exclusion Criteria:

* Previous treatment.
* Other ophthalmic diseases. history of Nephropathy, heart diseases and pregnancy
* Media opacities

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity

SECONDARY OUTCOMES:
Central Retinal Thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Eduarto Torres-Porras, MD, Study Director — Asociación para Evitar la Ceguera en México; Octavio Burgos, MD, Principal Investigator — Asociación para Evitar la Ceguera en México
Locations (1):
- Asociación para Evitar la Ceguera en México, Mexico City, Mexico City, Mexico